CLINICAL TRIAL: NCT05400486
Title: Comparison of the Additional Effects of Using TENS and Interferential Currents for the Treatment of Individuals With Chronic Nonspecific Neck Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Cid André Fidelis de Paula Gomes, Phd, professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 58624422.3.0000.5511
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Neck Pain; Chronic Pain
MeSH Terms: conditions — Neck Pain; Chronic Pain | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The principal investigator will not be part of any assessment or treatment process.
  Two researchers will be solely responsible for evaluating the outcomes. These will not participate in any other process. And they did not know the allocation of participants in their respective groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Therapeutic exercise group (Active Comparator): 1.Movements of flexion, extension, inclinations, and rotations of the cervical region at maximum amplitude and without load. 2.Neural mobilization of the cervical nerve roots. 3.Contraction of the deep muscles of the flexors, extensors, and rotators of the cervical region without performing spinal movements, using the movement of the eyes to aid in the accomplishment of these exercises. 4.Isometric contraction of the flexor muscles, inclinators, and rotators against manual resistance of the physiotherapist. 5.Isometric contraction of the cervical extensors of the cervical region against gravity. 6.Contraction of the flexor muscles, extensors, and incliners of the cervical region against the resistance of elastic bands.
  Interventions: Other: Therapeutic exercise
- Therapeutic exercise group + high frequency TENS (Experimental): This group will consist of 25 participants. Initially, TENS (Endophasys® - NMS-0501, KLD Biosistemas® Equipamentos Eletrônicos Ltda) will be applied to the cervical region through 4 silicon-carbon electrodes measuring 4 x 4 cm, with a water-based gel to reduce impedance at the skin-electrode interface. Thus, TENS will be applied with a rectangular, biphasic, and symmetrical pulse, with a pulse width of 100 µm, a frequency of 100 Hz, at the maximum tolerated sensitive threshold, for 30 minutes (VANCE et al., 2012). After the application of TENS, the same program of therapeutic exercises applied in the first group will be applied, in the same sequence, evolution, times, and repetitions.
  Interventions: Other: Therapeutic exercise; Other: Therapeutic exercise group + high frequency TENS
- Therapeutic exercise group + Interferential (Experimental): This group will consist of 25 participants. Initially, the protocol of exercises performed in the therapeutic exercise group will be applied. In sequence, the interferential current will be applied. Through the Endophasys® device - NMS-0501, KLD Biosistemas® Equipamentos Eletrônicos Ltda). Four electrodes (8x5 cm), two upper and two lower (forming a square) will be positioned around the center of the neck. The electrodes will be positioned crosswise, following the parameters: 4KHz (carrier frequency), 1/1 second (Sweep Mode), 60 Hz Amplitude of frequency modulation (AMF), 30 Hz (Delta AMF), automatic vector mode, with intensity at the motor threshold of sensation, lasting 30 minutes (Albornoz-Cabello et al., 2019).
  Interventions: Other: Therapeutic exercise; Other: Therapeutic exercise group + Interferential

INTERVENTIONS:
Other: Therapeutic exercise — 1.Movements of flexion, extension, inclinations, and rotations of the cervical region at maximum amplitude and without load. 2.Neural mobilization of the cervical nerve roots. 3.Contraction of the deep muscles of the flexors, extensors, and rotators of the cervical region without performing spinal movements, using the movement of the eyes to aid in the accomplishment of these exercises. 4.Isometric contraction of the flexor muscles, inclinators, and rotators against manual resistance of the physiotherapist. 5.Isometric contraction of the cervical extensors of the cervical region against gravity. 6.Contraction of the flexor muscles, extensors, and incliners of the cervical region against the resistance of elastic bands.
Other: Therapeutic exercise group + high frequency TENS — TENS (Endophasys® - NMS-0501, KLD Biosistemas® Equipamentos Eletrônicos Ltda) will be applied to the cervical region through 4 silicon-carbon electrodes measuring 4 x 4 cm, with a water-based gel to reduce the impedance at the interface electrode skin. Thus, TENS will be applied with a rectangular, biphasic, and symmetrical pulse, with a pulse width of 100 µm, and a frequency of 100 Hz, at the maximum tolerated sensitive threshold, for 30 minutes (VANCE et al., 2012).
  Arms: Therapeutic exercise group + high frequency TENS
Other: Therapeutic exercise group + Interferential — In sequence, the interferential current will be applied. Through the Endophasys® device - NMS-0501, KLD Biosistemas® Equipamentos Eletrônicos Ltda). Four electrodes (8x5 cm), two upper and two lower (forming a square) will be positioned around the center of the neck. The electrodes will be positioned crosswise, following the parameters: 4KHz (carrier frequency), 1/1 second (Sweep Mode), 60 Hz Amplitude of frequency modulation (AMF), 30 Hz (Delta AMF), automatic vector mode, with intensity at the motor threshold of sensation, lasting 30 minutes (Albornoz-Cabello et al., 2019).
  Arms: Therapeutic exercise group + Interferential

SUMMARY:
In the current clinical and scientific reality, conservative treatment is the most coherent clinical management with a view to the proper rehabilitation of patients with chronic neck pain, with a trend towards the use of therapeutic exercise. However, some uncertainty about the effectiveness of therapeutic exercises still remains, requiring further studies with high methodological rigor, especially with regard to multimodal treatment, such as the combination of therapeutic exercises with photobiomodulation. Thus, the objective of this project is to evaluate the effects of adding photobiomodulation to a program of specific therapeutic exercises for the treatment of individuals with chronic non-specific neck pain. To this end, 60 participants will be randomized into three groups: therapeutic exercise group + photobiomodulation (n = 20), and therapeutic exercise group. There will be 8 treatment sessions and participants will be evaluated before, after the 8 sessions, and 4 weeks after the end of treatment using the Numerical Pain Scale, Neck Disability Index, Catastrophic Thoughts about Pain Scale, and Tampa Kinesiophobia Scale. In the statistical analysis, a linear mixed model will be applied, considering the interaction between the time and group factors. Finally, the addition of photobiomodulation to a therapeutic exercise program is expected to generate clinical improvements for patients with chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

* With chronic neck pain (for more than 90 days)
* Identified according to the following criteria: NDI score ≥ 5
* Numerical Pain Scale (END) score ≥ 3 at rest or during active neck movement

Exclusion Criteria:

* Individuals who had a history of cervical trauma; head, face, or cervical surgery
* Degenerative diseases of the spine
* Pain radiating to the upper limbs
* Having been submitted to physiotherapeutic treatment for the cervical region in the last three months
* Use of analgesics, anti-inflammatory drugs, or muscle relaxants in the last week; the presence of systemic diseases
* medical diagnosis of fibromyalgia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2022-07-30 (Actual); Primary Completion 2025-04-20 (Actual); Study Completion 2025-04-20 (Actual)

PRIMARY OUTCOMES:
Functional disability | Change from Baseline after 8 weeks of intervention and 4 weeks after the end of the intervention.]
  The NDI will be used to verify the degree of disability due to neck pain.
Numerical Pain Scale | Change from Baseline after 8 weeks of intervention and 4 weeks after the end of the intervention.]
  The Numerical rating pain scale, a simple, easily administered scale evaluates the perceived intensity of pain, using an 11-point scale from 0, representing 'no pain', to 10, which is the 'worst possible pain'.

SECONDARY OUTCOMES:
Catastrophic Thoughts about Pain Scale | Change from Baseline after 8 weeks of intervention and 4 weeks after the end of the intervention.]
  The Catastrophic Thoughts About Pain Scale will be used to assess pain-related catastrophizing.
Kinesiophobia Tampa Scale | Change from Baseline after 8 weeks of intervention and 4 weeks after the end of the intervention.]
  Tampa Kinesiophobia Scale will be used to assess fear of movement and injury recurrence.
The Copenhagen Neck Functional Disability Scale (CNFDS) | Change from Baseline after 8 weeks of intervention and 4 weeks after the end of the intervention.]
  The CNFDS is a one-dimensional self-report scale consisting of 15 items that assess the degree of disability in activities of daily living in patients diagnosed with neck pain. When calculating the CNFDS score, the following procedures should be considered: For items 1 to 5, the answer "yes" = 0, "sometimes" = 1 and "no" = 2; For items 6 to 15, the answer "yes" = 2, "sometimes" = 1 and "no" = 0. Thus, the total score ranges from 0 to 30, the higher the score, the greater the disability.
Global Perception of Change Scale | Change from Baseline after 8 weeks of intervention and 4 weeks after the end of the intervention.]
  The perception of the global effect of the treatment by the research participant will be evaluated by the Global Perception of Change Scale. The Global Perception of Change Scale is a direct scale on the patient's self-perception when the intervention is performed. This scale is composed of 11 points, ranging from -5 (worse compared to the start of treatment), 0 (neutral) and +5 (improvement compared to the start of treatment), using the Portuguese version.

CONTACTS AND LOCATIONS:
Overall Officials: Cid Gomes, Phd, Principal Investigator — University of Nove de Julho
Locations (1):
- University of Nove de Julho, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
Make data available remotely in digital cloud storage.

REFERENCES:
- [Derived] de Santana GN, da Silva ACB, Dos Santos PG, Girasol CE, de Oliveira AR, Dibai-Filho AV, de Paula Gomes CAF. Does Adding Electroanalgesic Modalities to a Multimodal Therapeutic Program Improve Clinical Outcomes in Individuals With Chronic Nonspecific Neck Pain? A Randomised Controlled Trial. Eur J Pain. 2025 Oct;29(9):e70121. doi: 10.1002/ejp.70121. PMID 40910433